CLINICAL TRIAL: NCT05228782
Title: A Phase IIb 3 Arm Randomized Clinical Pilot Study to Assess the Impact of a Peer-support Program to Improve Social Isolation and Loneliness Due to COVID-19 - Comparing the Addition of a Secure, User Friendly Video-conference Solution and Telephone Support Alone to a Waiting List Control Group
Brief Title: COVID-19 and Social Isolation and Loneliness Trial
Acronym: SIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Bolton Clarke Research Institute (Unknown); Sunnybrook Research Institute (Other); North York General Hospital (Other); King's College London (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-0074E
Record Dates: First submitted 2021-10-01; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-09

CONDITIONS: Social Isolation; Loneliness; Geriatric
Keywords: Loneliness; Social Isolation; Emergency Department; Geriatrics; Geriatric Psychiatry; Family Medicine; Randomized Clinical Trial
MeSH Terms: conditions — Social Isolation; Emergencies

STUDY DESIGN:
Intervention Model Description: This multi-centered, three-arm, outcome assessor blinded randomized clinical trial will follow CONSORT reporting guidelines and is part of a program of research that adheres to the ORBIT model for developing complex behavioural interventions. In this model, the previous study by Lowthian and colleagues established the proof of concept, and the current trial Phase IIb is adequately powered to test whether two versions of the HOW R U? intervention are effective compared to a common standard care wait-list arm.
Who Masked: Outcomes Assessor
Masking Description: We will use intention-to-treat analysis for the primary outcome to further protect against selection bias. It is not feasible to blind participants to the intervention. Primary outcomes will be assessed after 12 weeks by a research assistant who has had no previous contact with participants and is blinded to the intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HOW RU Intervention delivered by telephone (Experimental): Group Phone will receive the HOW RU? intervention over the telephone.
  Interventions: Other: HOW R U? Intervention
- HOW RU Intervention delivered by video-call (Experimental): Group Video will receive the HOW RU? intervention delivered over video-call using the aTouch Away platform.
  Interventions: Other: HOW R U? Intervention
- Wait-list Control Group (No Intervention): Control groups will be offered standard care through their referring service (i.e. their routine clinical follow-up). The control group will be offered HOW RU? telephone support outside of the main trial after their primary outcome assessment at 12 weeks

INTERVENTIONS:
Other: HOW R U? Intervention — HOW RU? intervention uses trained volunteer peers to provide strength-based support sessions weekly for 12 weeks.
  Arms: HOW RU Intervention delivered by telephone; HOW RU Intervention delivered by video-call

SUMMARY:
Social isolation and loneliness worsen older peoples' quality of life, risk of dementia, and contributes to 45,000 deaths/year in Canada - as much as smoking. Isolated people use the health care system more often, but have worse outcomes. Effective, inexpensive interventions exist but unfortunately they have not been implemented in Canada.

We partnered with the Australian developer of HOW R U?, an effective and feasible intervention that uses specially trained, older, hospital volunteers to provide peer support to combat isolation and loneliness in isolated older peers.

Little is known about older people's preferences for virtual care (telephone vs. video) nor their relative effectiveness. Thus we will compare two ways of delivering HOW R U: telephone support and a tested, secure user-friendly video conferencing app, aTouch Away® to a common control arm.

We also partnered with Emergency Medicine, Family Medicine, Geriatrics and Psychiatry to identify people who will benefit from peer support; and with Volunteer Services to recruit volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Any community-dwelling person 70 years of age and older receiving care from the ED, Family Medicine, or Geriatric clinics at our two participating sites (MSH and NYGH) will be eligible.

Exclusion Criteria:

* age less than 70 years; communication problems (critically ill, unconscious, language barrier, speech impairment or otherwise unable to provide consent), or admission to a hospital for > 72 hours. Patients with severe cognitive impairment or those living in nursing homes who are dependent on others for their activity of daily living will be excluded. To target the intervention for older people with loneliness a baseline de Jonge loneliness scores of 2.0 will be required for participation in the trial.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-11-03 (Estimated)

PRIMARY OUTCOMES:
Change in De Jong Gierveld Loneliness Scale at Baseline | This scale will be collected at baseline and at 12 weeks.
  We will use the 6-item De Jong Gierveld loneliness scale as our primary outcome measure.The minimum value is 0 and the maximum value is 6.

SECONDARY OUTCOMES:
Change in Social Network | Baseline and at 12 weeks
  Lubben's Social Network Scale
Change in Mood | Baseline and at 12 weeks
  Geriatric Depression Scale
Change in Quality of life | Baseline and at 12 weeks
  EQ-5D-5L survey
all-cause mortality | Follow-up phone call at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lee JS, Rose L, Borgundvaag B, McLeod SL, Melady D, Mohindra R, Sinha SK, Wesson V, Wiesenfeld L, Kolker S, Kiss A, Lowthian J. Impact of a peer-support programme to improve loneliness and social isolation due to COVID-19: does adding a secure, user friendly video-conference solution work better than telephone support alone? Protocol for a three-arm randomised clinical trial. BMJ Open. 2024 Jan 9;14(1):e056839. doi: 10.1136/bmjopen-2021-056839. PMID 38199634